CLINICAL TRIAL: NCT07047742
Title: Assess the Efficacy of Dietary Interventions and Educational Programs as Adjunctive Therapies for the Management of Urolithiasis
Brief Title: Efficacy of Dietary Interventions and Educational Programs as Adjunctive Therapies for the Management of Urolithiasis: Efficacy of Fresh Lemon Juice and Roselle as Educational Program on Urolithiasis Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Dler Mohammed Saeed, Assistant lecturer, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2423
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Urolithiasis, Lemon Juice
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lemon juice group (Experimental): this group receive lemon juice as well as education about urolithiasis management as adjunctive therapy to their conventional treatments. the total participants of this group will be 50 participants.
  Interventions: Dietary Supplement: lemon juice; Other: Education on urolithiasis management
- Roselle group (Experimental): this group receive Roselle as well as education about urolithiasis management as adjunctive therapy to their conventional treatments. the total participants of this group will be 50 participants.
  Interventions: Dietary Supplement: Roselle; Other: Education on urolithiasis management
- education (Experimental): this group receive only education about urolithiasis management as adjunctive therapy to their conventional treatments. the total participants of this group will be 50 participants.
  Interventions: Other: Education on urolithiasis management
- control group (No Intervention): this group is a control group. they receive no intervention and just receive their coventional treatment. the total participants of this group will be 50 participants.

INTERVENTIONS:
Dietary Supplement: lemon juice — in this study for the first arm fresh lemon juice two times daily is advised
  Arms: lemon juice group
Dietary Supplement: Roselle — for the second arm Roselle tea is advised tow times per day
  Arms: Roselle group
Other: Education on urolithiasis management — all the arms except control group receive education about urolithiasis management
  Arms: Roselle group; education; lemon juice group

SUMMARY:
The Efficacy of Dietary and Health Educational Program, as Adjunctive Therapies for the Management of Urolithiasis Introduction Background Urolithiasis, commonly known as kidney stone disease, is a prevalent global health concern affecting millions of individuals annually. The incidence and recurrence of urolithiasis have been increasing due to dietary habits, metabolic disorders, and genetic predispositions (Qian et al., 2022). Kidney stones are crystalline mineral deposits that form within the urinary tract and are classified based on their chemical composition, including calcium oxalate, uric acid, struvite, and cystine stones (Wang et al., 2021).The condition is associated with debilitating symptoms such as renal colic, hematuria, and urinary tract obstruction, leading to significant morbidity and healthcare costs (Urolithiasis EAU Guidelines on, 2023).Conventional management strategies for urolithiasis include pharmacological treatments, extracorporeal shock wave lithotripsy (ESWL), ureteroscopy, and surgical interventions (Fedorowicz et al., 2024). Despite these treatments, high recurrence rates highlight the necessity of preventive strategies through dietary and lifestyle modifications.

Complementary and alternative medicine (CAM) has gained increasing attention in urolithiasis prevention and management, particularly the use of herbal remedies and nutritional interventions. Citrus fruits, particularly lemon juice, have been proposed as effective dietary interventions due to their high citrate content, which inhibits stone formation (Ruggenenti et al., 2022). Additionally, Hibiscus sabdariffa (roselle) has been traditionally used for its diuretic and nephroprotective properties, suggesting potential benefits in preventing urolithiasis (Prasongwatana et al., 2018). However, while these natural interventions have shown promise, there is a lack of strong clinical evidence supporting their efficacy in reducing kidney stone formation and recurrence. Additionally, patient education is crucial in modifying lifestyle behaviors and improving adherence to preventive measures (Gamal et al., 2023). Thus, a comprehensive approach integrating dietary interventions with structured education could be more effective in managing urolithiasis.

Aim of study This study aims to evaluate the efficacy of dietary interventions (fresh lemon juice and Hibiscus sabdariffa) combined with an educational program in managing urolithiasis.

Objectives of study

This dissertation has several objectives which are listed below:

1. Evaluate the effectiveness of fresh lemon juice, in conjunction with an educational program, on the urinary stones parameters (like stone size, symptoms, infection rate, …), as well as tracking its potential complications.
2. Evaluate the effectiveness of Hibiscus sabdariffa (Roselle) in conjunction with an educational program, on the urinary stones parameters (like stone size, symptoms, infection rate, …), as well as tracking its potential complications.
3. To determine the effectiveness of educational program on the urinary stones parameters (like stone size, symptoms, infection rate, …)
4. To compare the outcomes among four study groups: (i) lemon juice + education, (ii) roselle tea + education, (iii) education-only, and (iv) control (no intervention).
5. Assess demographic data and clinical status, stone characteristics, lifestyle and dietary habits of participants.
6. Assess knowledge and attitude of participants regarding complementary and alternative medicine (CAM).

DETAILED DESCRIPTION:
Study Design

This study employ a prospective, randomized controlled trial (RCT) design to evaluate the efficacy of dietary interventions-fresh lemon juice and hibiscus sabdariffa (Roselle)-combined with structured education, as adjunctive therapies to conventional treatments for urolithiasis management. The study comprise four parallel groups, each consisting of 50 participants, randomized into the following groups:

1. Lemon Juice + Education Group Received 30-60 mL of fresh lemon juice twice daily alongside a standardized educational program.
2. Roselle + Education Group Administered 1.5 g of hibiscus sabdariffa tea twice daily with the same educational intervention.
3. Education-Only Group Provide solely with the educational program.
4. Control Group Receive no dietary intervention or education, continuing conventional treatments as prescribed.

The trial duration lasts 12 weeks, with follow-up assessments at 4-week intervals (4th, 8th, and 12th weeks) to monitor adherence, symptom progression, and urinary stone parameters. Randomization was stratified by age and gender to ensure balanced group allocation.

Study Setting

The study is conduct in three hospitals in Erbil governorate in the Kurdistan region of Iraq:

* Shaqlawa Teaching Hospital
* Pirmam Teaching Hospital
* Rizgary Teaching Hospital These hospitals will be selected based on their patient population, availability of diagnostic facilities, and accessibility for follow-up assessments. Each hospital has specialized urology units and laboratories capable of conducting the required tests, ensuring consistency in data collection.

Data Collection The intervention phase, lasting approximately three to four months, represented the core data collection stage of my study. During this period, I actively visit selected hospitals to recruit participants, ensuring that the study met the required sample size while maintaining methodological rigor.

Based on my sample size calculations, I initially aimed to recruit at least 200 participants, who were then randomly assigned into four groups:

1. Lemon juice + education
2. Roselle + education
3. Education only
4. Control (no intervention)

Follow-up and Schedule

Participants will followed up at four key time points:

* Baseline (Week 0) Initial assessment, which include completing study questionnaire including demographic data, clinical history, dietary habits, life style, knowledge and attitude regarding complementary and alternative medicine (CAM) and urolithiasis parameters (urinalysis and ultrasound).
* First follow up (Week 4) First follow-up to assess dietary adherence, symptom changes, side effects and urolithiasis parameters (urinalysis and ultrasound).
* Second Follow up (Week 8) Midpoint follow-up for further evaluation of intervention effectiveness which include dietary adherence, symptom changes, side effects and urolithiasis parameters (urinalysis and ultrasound).
* Third Follow up (Week 12) Final follow-up to determine long-term changes in urolithiasis characteristics and overall outcomes, which include dietary adherence, symptom changes, side effects and urolithiasis parameters (urinalysis and ultrasound), as well as asking some questions about attitude of participants regarding CAM (the same questions asked from the participant at the baseline assessment) to track and identify changes in their attitude regarding CAM through this period.

Throughout the follow-up period, I will maintain direct contact with participants to ensure adherence and minimize dropouts.

Data Entry and Analysis The data entry and analysis phase, spanning two months, is a critical stage in the study, ensuring that collected data is accurately recorded, processed, and interpreted. During this period, all completed questionnaires, urinalysis reports, and ultrasound findings will be systematically entered into SPSS software to create a structured database for statistical analysis. Data cleaning conducted to identify and correct errors, such as missing values or inconsistencies, ensuring the dataset is reliable and ready for interpretation. Following this, statistical tests will be performed to assess the impact of the dietary interventions and educational program on urolithiasis outcomes, comparing the results across study groups. This step involves both descriptive and inferential statistical methods, such as t-tests, ANOVA, or regression analysis, depending on the nature of the variables and research objectives. The findings are summarized into tables and figures to facilitate interpretation and presentation in the dissertation. As this phase directly influences the validity of study conclusions, meticulous attention is given to accuracy, consistency, and adherence to statistical assumptions.

Participants and Sampling Target Population The target population for this study consists of individuals diagnosed with urolithiasis in Erbil governorate, Iraq, who seek medical care at Shaqlawa, Pirmam, and Rizgary hospitals. These participants represent a diverse demographic group with varying risk factors, dietary habits, and lifestyle behaviors that may influence the development and management of kidney stones.

Inclusion Criteria

The following aspects is considered for the inclusion of participants in the study:

* Adults aged 18-75 years diagnosed with urolithiasis.
* Patients are willing to participate and provide informed consent.
* Patients do not currently use lemon juice, Roselle, or other herbal treatments for urolithiasis.
* No history of severe gastrointestinal disorders or metabolic conditions interfering with dietary interventions.

Exclusion Criteria

Based on predefined criteria, patients excluded if they have:

* Allergies to citrus fruits or hibiscus.
* Chronic kidney disease (CKD) stage 3 or higher.
* Pregnancy or lactation.
* Gastrointestinal disorders (e.g., GERD, ulcers, chronic gastritis for lemon juice group).
* Metabolic disorders (e.g., hyperparathyroidism, gout, hyperoxaluria).
* Recent urolithiasis surgery (within the last 3-6 months).
* Severe systemic diseases (e.g., cancer, advanced cardiovascular diseases).
* Hypertension requires diuretics (due to potential interaction (synergic effect) between dietary interactions and prescribed medications for hypertension which may lead to hypotension).
* Malabsorption disorders (e.g., Crohn's disease, celiac disease).
* Non-compliance with study protocols. The exclusion criteria ensure homogeneity in the study sample and improve the reliability of intervention assessment.

Sample Size Calculation Sample size was determined using G Power software, setting α = 0.05 and power = 0.80, as a common standard for most research resulting in 50 participants per group, for a total of 200 participants. I selected an effect size of 0.25, which is commonly considered moderate effect size for sample calculation with G power program. It means that lemon juice or Roselle moderately affect urinary stone parameters. Power analysis ensures sufficient sensitivity to detect meaningful differences between intervention and control groups.

Sampling Method A consecutive sampling strategy will be employed, enrolling eligible patients from outpatient urology consultation clinics. It means that every eligible participant who meets the inclusion criteria is systematically recruited until the required sample size is reached. Participants are screened based on their medical history, urinalysis, and ultrasound results to confirm the presence of kidney stones. Eligible individuals who provide informed consent are then assigned to one of four groups, each containing 50 participants: (1) lemon juice + education, (2) roselle + education, (3) education only, and (4) control (no intervention).

Randomization Process To ensure the validity of comparisons between study groups and minimize potential confounding factors, participants randomly assigned to one of the four groups after enrollment. Block randomization is used to achieve a balanced distribution of participants across the groups, ensuring that each group receives an equal number of participants. Blocks of fixed or variable sizes (e.g., 4 or 8 participants per block) are generated, and participants are assigned using a computer-generated randomization list. This method helps prevent imbalances in baseline characteristics, such as age, gender, or stone type, across the groups. The allocation sequence is concealed until the moment of assignment to reduce selection bias. Since the nature of the interventions (lemon juice, roselle, education) makes blinding difficult, the study follows an open-label design, where participants and researchers are aware of the assigned interventions. However, outcome assessors analyzing urinalysis and ultrasound results remain blinded to the intervention groups to minimize assessment bias. This randomization process ensures that differences in outcomes are attributable to the interventions rather than systematic differences between groups.

Research Ethics This study adheres to strict ethical guidelines to ensure the rights, safety, and well-being of all participants. Ethical approval was obtained from the Hawler Medical University ethics committee (Reference number: 2423) before initiating the study, ensuring compliance with national and international research standards (Appendix 1). Additionally, administrative permissions were secured from Shaqlawa, Pirmam, and Rizgary hospitals in Erbil governorate, Iraq, where participant recruitment took place, after initial approval from directorate of health.

All participants provide written informed consent before enrollment, confirming their voluntary participation and understanding of the study objectives, procedures, potential benefits, and risks. The informed consent formed will be translated to Kurdish language which is the native language of the area, and asked participants to carefully read and sign it after taking full information about the study from researcher. They informed that they had the right to withdraw from the study at any time without any consequences for their medical care. Confidentiality and anonymity strictly maintained by assigning unique identification codes instead of using personal information in data records. All data securely stored and accessible only to authorized research personnel.

Additionally, special attention will be given to scientific integrity and data transparency, ensuring that findings were reported accurately without fabrication or manipulation. By upholding these ethical standards, the study guarantees participant protection, data integrity, and adherence to ethical research principles in evaluating the efficacy of dietary and educational interventions for urolithiasis management.

Interventions of the Study Dietary Interventions The study involves two dietary interventions, fresh lemon juice and Hibiscus sabdariffa (roselle) tea, which are provided alongside conventional treatments for urolithiasis. These interventions aim to assess their effectiveness in reducing urinary stone formation, improving symptoms and outcomes, and modifying urinary parameters. More description about each interventional group is discussed below.

A. Lemon Juice Group Participants in this group consume 30-45 ml (one average size citrus lemon) of freshly squeezed lemon juice twice daily, preferably after meals, with a full glass of water to enhance absorption and minimize gastrointestinal discomfort and enamel erosion. The participants are instructed to dilute the lemon juice in water to prevent potential dental enamel erosion from citric acid. Compliance and complications is monitored through follow-up interviews at 4, 8, and 12 weeks to evaluate adherence and effectiveness.

B. Roselle (Hibiscus sabdariffa) Group Participants in this group will be instructed to consume 1.5 g of dried grinded Hibiscus sabdariffa in the form of tea, prepared by pouring 1 teaspoon dried flowers in 100 to 150 ml of hot water for 5-10 minutes. This tea is consumed twice daily. Because of lack of knowledge about this material among the population and to decreased costs burden of preparing it for the participants, this material is prepared for the participants by researcher. Average cost of one kilogram of Roselle dry calyces in Erbil is approximately 8 - 10 $, which is inexpensive into some extent. Roselle dried calyces are moderately grinded and offered to the participants in a package which was enough to cover intervention duration (12 weeks). A premeasured teaspoon which could carry 1.5 gram of Roselle with each use provides a meticulously right dose for this intervention. Participants were fully educated about the method of drinking Roselle tea and advised to avoid adding excess sugar to the tea. Compliance and complications is tracked through follow-up assessments at 4, 8, and 12 weeks.

Educational Program The educational program is an integral part of the intervention for the Lemon Juice, Roselle, and Education-Only groups. This program is designed to increase participants' knowledge about urolithiasis and provide actionable guidance on managing and preventing kidney stones through dietary and lifestyle modifications. Because gathering all the participants may not applicable each participant individually educate by researcher and after finishing the education process a handout which summarizes important points of education program (which will be translated to native participant language) is offered to the participant.

To assess the effectiveness of the dietary and lifestyle interventions, the program includes regular monitoring and follow-up. Participants will be encouraged to adhere to schedule regular follow-up visits to monitor their condition using ultrasound and urine analysis to track the size, number, and type of kidney stones. This helps assess any changes in urinary parameters and provides early detection of potential complications. Participants are advised to report any changes in symptoms during their visits.

The program includes a series of structured educational sessions that cover various aspects of urolithiasis, as outlined below.

1. Introduction to Urolithiasis

   * Definition and Prevalence: Urolithiasis refers to the formation of stones in the urinary tract, which can cause pain and lead to urinary issues. Common types of kidney stones include calcium oxalate, uric acid, and struvite stones.
   * Risk Factors: The educational program highlights risk factors that contribute to kidney stone formation, such as dehydration, high salt intake, high-protein diet, obesity, and other medical conditions that increase the likelihood of stone formation.
2. General Health Education

   * Hydration

     * Importance of Hydration: Maintaining proper hydration helps dilute the substances in urine that can form stones.
     * Recommendation: Participants are encouraged to drink at least 2-3 liters of water daily (about 8-12 glasses), which helps flush out minerals and prevents them from crystallizing into stones.
   * Dietary Changes

     * Reduce Salt Intake: High salt intake can lead to increased calcium in the urine, which promotes stone formation. Participants are advised to consume less than 2,300 milligrams of sodium per day (equivalent to 1 teaspoon of salt).
     * Balanced Diet: A diet rich in fruits and vegetables helps reduce the risk of kidney stones by increasing urinary citrate levels, which act as inhibitors for stone formation.
     * Adequate Calcium Intake: Participants are instructed to ensure an adequate intake of calcium (1,000-1,200 mg daily) through dietary sources like dairy products, leafy greens, and fortified foods. Low calcium intake can lead to increased oxalate absorption.
     * Limit Animal Protein: High intake of animal protein (e.g., meat, fish, and poultry) increases the risk of stone formation. The program recommends limiting these foods to 0.8-1 g per kg body weight per day.
     * Avoid Oxalate-Rich Foods: Foods high in oxalates (such as spinach, rhubarb, beets, nuts, especially almonds and cashews, chocolate, and black tea) can contribute to stone formation. Participants are advised to limit these foods if prone to oxalate stones.
   * Lifestyle Modifications

     * Exercise: Regular physical activity helps maintain a healthy weight and reduces the risk of kidney stone formation. Participants are encouraged to aim for at least 150 minutes of moderate-intensity exercise per week.
     * Avoid Sugary Drinks: Sugary beverages are associated with an increased risk of kidney stones, and participants are encouraged to limit or avoid them, opting for water, herbal teas, or other non-sugary drinks.
     * Limit Alcohol Consumption: Excessive alcohol consumption can lead to dehydration, which increases the risk of stone formation. The program advises participants to limit their alcohol intake.

Data Collection Instruments Study Questionnaire The study questionnaire meticulously designed to collect comprehensive data on participants' socioeconomic profiles, medical and surgical histories, dietary and lifestyle habits, knowledge and attitudes toward complementary therapies, and clinical outcomes related to urolithiasis. Developed through an iterative process involving expert consultations and pilot testing, the instrument integrates both quantitative and qualitative elements to capture multifaceted insights into the efficacy of dietary interventions and education. Below is a detailed breakdown of its structure and components.

1. Questionnaire Structure The questionnaire comprises eight distinct sections, each targeting specific domains relevant to the study's objectives. I completed the questionnaire through direct interviews with the patients to ensure that all terms and questions were fully understood. This approach allows for clarification of any doubts or confusion, ensuring accurate and meaningful responses. Additionally, conducting interviews in person helps to establish rapport and ensures that the patient feels comfortable, which can lead to more reliable data. By interacting directly with the participants, I can also observe non-verbal cues and ensure that all aspects of the questionnaire are addressed thoroughly. Different parts of the questionnaire is briefly discussed below.

   1.1. Socioeconomic Data (Part I)

   This section gathers foundational demographic information to contextualize participants' backgrounds:

   • Age: Recorded in years to analyze age-related trends in intervention efficacy.
   * Gender: Categorized as male or female to explore gender-specific responses.
   * Occupation: Options include employed, unemployed, housewife, retired, or "other" with a free-text field for specificity.
   * Education Level: Ranges from illiteracy to university graduation, assessing potential correlations between education and health literacy.
   * Marital Status: Includes single, married, widowed, or divorced to evaluate social support influences.
   * Income Level: Stratified as high, moderate, or low to examine socioeconomic impacts on dietary adherence.
   * Anthropometrics: Height, weight, and BMI measurements provide baseline health metrics.

   1.2. Medical History (Part II)

   This segment investigates participants' clinical backgrounds:
   * Kidney Stone History: Documents prior diagnoses, duration, stone type (e.g., calcium oxalate, uric acid), and current symptoms (e.g., colic, hematuria).
   * Chronic Conditions: Checklists for hypertension, diabetes, and cardiovascular diseases identify comorbidities that may influence outcomes.
   * Medication Use: Open-ended questions list prescribed drugs to assess interactions with interventions and main types of conventional medications which mainly used to treat urolithiasis.
   * Family History: Identifies genetic predispositions to urolithiasis. 1.3. Surgical History (Part III) Participants report prior stone-related surgeries (e.g., ESWL, PCNL) to control procedural impacts on stone recurrence or intervention response.

   1.4. Dietary Habits (Part IV)

   A detailed exploration of nutritional patterns includes:
   * Fluid Intake: Daily water consumption (mL) and frequency of sugary/cola beverages.
   * Salt and Meat Consumption: Likert-scale items quantify intake of processed foods and animal protein.
   * Dairy and Citrus Use: Frequency of dairy products, lemon juice, and hibiscus tea consumption, critical for evaluating level of consumption among participants.

   1.5. Lifestyle (Part V)

   This section assesses modifiable risk factors:

   • Physical Activity: Categorized as low, moderate, or high to gauge exercise's role in stone prevention.
   * Substance Use: Smoking habits (type, frequency) and alcohol consumption patterns.
   * Stress Management: Multiple-choice responses (e.g., exercise, meditation) identify coping mechanisms affecting overall health.

   1.6. Knowledge of Complementary Therapies (Part VI)

   Multiple-choice and Likert-scale questions evaluate participants' understanding of herbal medicine's role, including:
   * Purpose of Complementary Therapies: Distinguishes between replacement vs. adjunctive use.
   * Herbal Medicine Principles: Tests knowledge of plant-based healing versus synthetic alternatives.
   * Information Sources: Identifies whether participants rely on healthcare providers, family, or online resources for herbal advice.

   1.7. Attitude Toward Complementary Therapies (Part VII)

   Administered at baseline and 12-week follow-up, this section uses a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree) to measure shifts in perceptions, such as:

   • Efficacy of herbal remedies in stone management.
   * Preference for integrating complementary therapies with conventional treatments.
   * Concerns about self-treatment risks. 1.8. Follow-Up Assessments (Part VIII)

   Structured interviews at 4, 8, and 12 weeks track:

   • Adherence: Binary (yes/no) questions confirm compliance with lemon juice, hibiscus, or education protocols.
   * Symptom Changes: Open-ended descriptions of pain, dysuria, or hematuria progression.
   * Side Effects and Barriers: Free-text fields document adverse reactions (e.g., gastrointestinal discomfort) or challenges (e.g., taste aversion).
   * Pain Severity: Numeric rating scales (1-10) quantify subjective pain levels.
   * Lab/Ultrasound Data: Structured tables record objective metrics (stone size, location, counts and urinary parameters) across follow-ups.

   Validation and Reliability

   To ensure robustness, the questionnaire underwent rigorous validation:

   • Content Validity: Questionnaire was reviewed by 10 experts in the field of adult nursing. They reviewed the instrument for relevance and clarity to achieving content validity.
   * Pilot Testing: 10 participants recruit two times to complete the questionnaire with two weeks interval after first intervention time. Test-retest reliability analysis revealed strong consistency (I will write the test result later).
   * Internal Consistency: Cronbach's α for Likert-scale sections ranged (I will write the test result later), indicating high reliability.

   Clinical and Laboratory Assessments

   Participants undergo the following clinical and laboratory assessments as well as completing the questionnaire. They briefly listed below:

   • Urinalysis (RBCs, pus cells, pH, crystals, bacteria)
   * Ultrasound (number, size, and location of stones)
   * Anthropometric measures: Height, weight, BMI Assessments occur at baseline, 4 weeks, 8 weeks, and 12 weeks after initial visit."

ELIGIBILITY:
Inclusion Criteria:

* The following aspects is considered for the inclusion of participants in the study:

  * Adults aged 18-75 years diagnosed with urolithiasis.
  * Patients are willing to participate and provide informed consent.
  * Patients do not currently use lemon juice, Roselle, or other herbal treatments for urolithiasis.
  * No history of severe gastrointestinal disorders or metabolic conditions interfering with dietary interventions.

Exclusion Criteria:

* Based on predefined criteria, patients are excluded if they have:

  * Allergies to citrus fruits or hibiscus.
  * Chronic kidney disease (CKD) stage 3 or higher.
  * Pregnancy or lactation.
  * Gastrointestinal disorders (e.g., GERD, ulcers, chronic gastritis for lemon juice group).
  * Metabolic disorders (e.g., hyperparathyroidism, gout, hyperoxaluria).
  * Recent urolithiasis surgery (within the last 3-6 months).
  * Severe systemic diseases (e.g., cancer, advanced cardiovascular diseases).
  * Hypertension requires diuretics (due to potential interaction (synergic effect) between dietary interactions and prescribed medications for hypertension which may lead to hypotension).
  * Malabsorption disorders (e.g., Crohn's disease, celiac disease).
  * Non-compliance with study protocols. The exclusion criteria ensure homogeneity in the study sample and improve the reliability of intervention assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in kidney stone size measured by ultrasound | Baseline and 12 weeks after intervention
  Change in the largest diameter (in mm) of kidney or ureteral stones as measured by abdominal ultrasound.

SECONDARY OUTCOMES:
Change in participant attitude score regarding complementary alternative medicine (CAM) | Baseline and 12 weeks
  Assessed using a structured questionnaire, scored and compared from baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Rizgary teaching Hospital, Pirmam teaching hospital, Shaqlawa teaching hospital, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to participant privacy concerns and local ethical approval limitations.